CLINICAL TRIAL: NCT05331482
Title: Effectiveness of Two Exercise Programs on the Neck. Secondary Analysis of a Randomized Clinical Trial.
Brief Title: Effectiveness of Two Exercise Programs on the Neck.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Pilar Pardos Aguilella, Colaborator Lecturer in Physiotherapy, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.P.-C.I.PI21/357
Record Dates: First submitted 2022-04-10; First posted 2022-04-15 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2023-08

CONDITIONS: Subjects With Deep Cervical Muscle Strength Deficit
Keywords: neck muscles; neck pain; exercise therapy; telerehabilitation; muscle weakness
MeSH Terms: conditions — Neck Pain; Muscle Weakness | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial with 3 different groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Training protocol with the cervical device for treatment (CDAT). (Experimental): Endurance training program of deep cervical flexors and deep cervical extensors with the cervical device for treatment.
  Interventions: Other: Training protocol with the cervical device for treatment (CDAT).
- Conventional training protocol- (Active Comparator): Endurance training program of deep cervical flexors and deep cervical extensors with the conventional protocol.
  Interventions: Other: Conventional training protocol
- Control Group (No Intervention): Subject continues with activities of daily living. Does not receive deep cervical muscle training.

INTERVENTIONS:
Other: Training protocol with the cervical device for treatment (CDAT). — Endurance training program of deep cervical flexors and deep cervical extensors with the cervical device for treatment.
  Arms: Training protocol with the cervical device for treatment (CDAT).
Other: Conventional training protocol — Endurance training program of deep cervical flexors and deep cervical extensors with conventional training protocol.
  Arms: Conventional training protocol-

SUMMARY:
The purpose of this study is to evaluate the clinical results in lower cervical range of motion, size deep muscles, endurance, craniovertebral angle and cervical propioception by a training protocol with the new device for cervical treatment (CDAT) and the conventional training protocol (CT) versus a control group (C) in subjects with cervical deep muscle strength deficit.

DETAILED DESCRIPTION:
Neck pain is one of the major public health problems, which has a great impact on people's lives, with high prevalence and recurrence rate. Cervical vertebral column is heavily dependent on the muscles for its physical support and activities. There are increasing evidences to support that cervical muscles may impair in patients with neck disorders. Training protocols can help to improve pain, cervical function, posture and cross-sectional area. However, there are no training protocols in subjects with strength deficit of deep cervical muscles, including deep neck extensor and flexor muscles. The cervical device treatment (CDAT) allows us to train the cervical flexor and extensor muscle in a simple and comfortable way.

ELIGIBILITY:
Inclusion Criteria:

* Deep flexor strength deficit in craniocervical flexion test.
* Deep extensor strength deficit in neck extensor muscle endurance.
* ≤ 14 score in Neck disability Index

Exclusion Criteria:

* Have received cervical treatment during the last six month, presented any red flag, neurological or cognitive impairment (inability to understand the questionnaires or examination).
* Have received cervical manual therapy treatment during the last six month.
* A history of cervical trauma or surgery during the last year.
* Chronic neck pain occurring during the last six months (intensity, visual analogue scale >3/10, frequency > 2 days/week, duration >3 hours/day).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Deep neck flexor endurance Test. | Baseline and 6 weeks, 10 weeks, 14 weeks
  The Chin Tuck Neck Flexion Test is an assessment technique intended to determine the endurance of the deep cervical flexors.
Neck extensor muscle endurance Test | Baseline and 6 weeks, 10 weeks, 14 weeks
  Mean change from baseline in neck extensor muscle endurance Test after 6 weeks, 10 weeks and 14 weeks. The examiners assess the endurance of deep cervical extensor muscle.
Measurement of Cervical Multifidus and Longus Colli Muscle size. | Baseline and 6 weeks, 10 weeks, 14 weeks
  The examiners assess these deep muscles with ultrasound after 6 weeks, 10 weeks and 14 weeks.
Physical activity enjoyment Scale (PACES) | 6 weeks
  The examiners assess participant satisfaction with cervical deep muscle training.
  This scale measures enjoyment during physical activity through 16 items, which are preceded by the phrase "When I am active..." This instrument measures enjoyment and bipolar enjoyment, through statements such as "I enjoy it", "I'm bored", "It's very exciting", and "I don't like it". The answers will be collected on a Likert scale from 1 (totally disagree) to 5 (totally agree).

SECONDARY OUTCOMES:
Neck Disability Index | Baseline and 6 weeks, 10 weeks, 14 weeks
  Mean change from baseline in Neck Disability Index (NDI) (Neck Function) after 6 weeks , 10 weeks and 14 weeks.
  The examiners assess the self-perceived disability from neck pain using the NDI. The Neck Disability Index (NDI) is designed to measure neck-specific disability. The questionnaire has 10 items concerning pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation. The measure is designed to be given to the patient to complete.
  Item scores range from 0 (no disability) to 5 (total disability), with the minimum score is 0 (no disability) and maximum score of 50 (complete disability).
Neck Pain | Baseline and 6 weeks, 10 weeks, 14 weeks
  Mean change from baseline in neck pain (VAS) after 6 weeks, 10 weeks and 14 weeks. The examiners assess the self-perceived intensity of neck pain using the Visual Analogue Scale (VAS). The VAS is designed to measure pain intensity. It consists of a 10 cm horizontal line where the patient marks the point that best represents their pain, ranging from 0 (no pain) to 10 (worst imaginable pain). The measure is designed to be completed directly by the patient. Scores are recorded in centimeters, with higher values indicating greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Pardos-Aguilella, Principal Investigator — UicCatalunya
Locations (1):
- Élite Fisioterapia, María Montessori 2., Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No